CLINICAL TRIAL: NCT01347307
Title: Phase IV Trial Evaluating the Use of Stereotactic Body Radiotherapy for the Treatment of Spine Metastases and Primary Spine Tumors
Brief Title: Stereotactic Body Radiotherapy for Spine Tumors
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Mercy Research (Other)
Responsible Party: Principal Investigator, Juli Mai, MD, Radiation Oncology, Mercy Research
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 08-044
Record Dates: First submitted 2011-05-02; First posted 2011-05-04 (Estimated); Results first posted 2020-06-18 (Actual); Last update posted 2020-06-18 (Actual); Status verified 2020-06

CONDITIONS: Spinal Metastases; Vertebral Metastases; Benign Spinal Tumors; Chordoma; Meningioma; Schwannoma; Neurofibroma; Paragangliomas; Arteriovenous Malformations
Keywords: stereotactic radiotherapy; spinal metastases; vertebral metastases; benign spinal tumors
MeSH Terms: conditions — Chordoma; Meningioma; Neurilemmoma; Neurofibroma; Paraganglioma; Arteriovenous Malformations | interventions — Radiosurgery

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- SBRT for Benign Extradural Spine Tumors (Other): Benign extradural spine tumors such as chordomas, meningiomas, schwannomas, neurofibromas, paragangliomas, and arteriovenous malformations (AVMs).
  Interventions: Radiation: SBRT for Benign Extradural Spine Tumors
- SBRT for Vertebral/Paraspinal Metastases (Other): Vertebral and/or paraspinal metastases, with or without prior surgery and/or fractionated radiotherapy
  Interventions: Radiation: SBRT for Vertebral/Paraspinal Metastases

INTERVENTIONS:
Radiation: SBRT for Benign Extradural Spine Tumors — 14-25 Gy / 1 fraction OR 21-27 Gy / 3 fractions (7-9 Gy per fraction) OR 25-30 Gy / 5 fractions (5-6 Gy per fraction)
  Other Names: Stereotactic Body Radiotherapy (SBRT)
  Arms: SBRT for Benign Extradural Spine Tumors
Radiation: SBRT for Vertebral/Paraspinal Metastases — 12-16 Gy / 1 fraction OR 21-27 Gy / 3 fractions (7-9 Gy per fraction) OR 25-30 Gy / 5 fractions (5-6 Gy per fraction)
  Other Names: Stereotactic Body Radiotherapy (SBRT)
  Arms: SBRT for Vertebral/Paraspinal Metastases

SUMMARY:
This study will evaluate the local control rate as well as acute and late toxicity rates of stereotactic body radiotherapy (SBRT) for the treatment of spine metastases and benign spine tumors.

DETAILED DESCRIPTION:
This study is a single site, non-randomized, prospective, phase IV trial. Patients are composed of 2 groups:Spine Metastases OR Benign Spine Tumors. Data collected will include patient demographics, pathology data, tumor stage, SBRT dose fractionation scheme, dose received by adjacent critical normal tissues, tumor recurrence data, and acute and late toxicities.

Follow up data will be collected during the patient's standard office visits. The anticipated duration of this study is 5 years

ELIGIBILITY:
Eligibility Criteria:

* Patient age >= 18 years
* performance status of 0-3
* Vertebral and/or paraspinal metastases, with or without prior surgery and/or fractionated radiotherapy
* Benign extradural spine tumors such as chordomas, meningiomas, schwannomas, neurofibromas, paragangliomas, and arteriovenous malformations (AVMs).
* Established histologic diagnosis of a benign or malignant tumor of the spine.
* Arteriovenous malformation of the spine identified radiographically (no biopsy)
* Well-defined lesion involving no more than 2 adjacent vertebral levels or spinal segment
* Minimal spinal canal compromise that is not rapidly progressive. Ideally, the tumor should not be within 5 mm of the spinal cord.
* If chemotherapy is planned, ideally it should not have been given within 30 days of starting radiation and should not resume until at least 2 weeks after completing radiation. In addition, it is not recommended to perform SBRT when targeted anti-angiogenesis therapy is planned within 2 months of the procedure.
* Signed study-specific consent form

Exclusion Criteria:

* Lesion involving > 3 adjacent vertebral levels
* Overt spinal instability
* Neurologic deficit due to bony fragments/bony compression of neural structures
* Prior radiotherapy at the involved level(s) within 3 months of radiosurgery, more than one prior course of radiotherapy at the involved level(s), or more than 45 Gy previous radiation exposure at the involved level(s)
* Rapidly progressive spinal cord compromise or neurological deficit
* Paralysis, or otherwise compromised motor function due to radiographically confirmed cord compression
* Patient unable to undergo an MRI
* Pregnant or lactating women, due to potential exposure of the fetus to RT and unknown effects of RT on lactating females
* Patients with psychiatric or addictive disorder that would preclude obtaining informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 38 (Actual)
Dates: Start 2008-09 (Actual); Primary Completion 2017-09 (Actual); Study Completion 2017-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Bethany Sleckman, MD, Study Chair — Mercy Research
Locations (1):
- Mercy Medical Center, St. Louis, St Louis, Missouri, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- SBRT for Benign Extradural Spine Tumors: Benign extradural spine tumors such as chordomas, meningiomas, schwannomas, neurofibromas, paragangliomas, and arteriovenous malformations (AVMs).
  Stereotactic Body Radiation Therapy (SBRT) for Benign Extradural Spine Tumors: 14-25 Gy / 1 fraction OR 21-27 Gy / 3 fractions (7-9 Gy per fraction) OR 25-30 Gy / 5 fractions (5-6 Gy per fraction)
Period: Overall Study
Arm/Group | SBRT for Benign Extradural Spine Tumors | SBRT for Vertebral/Paraspinal Metastases
Started | 3 | 33
Completed | 3 | 28
Not Completed | 0 | 5
Not completed — Death | 0 | 4
Not completed — Physician Decision | 0 | 1

BASELINE CHARACTERISTICS:
Population: 2 enrolled patients were not treated. 35 patients completed 36 Stereotactic Body Radiotherapy courses for a total of 38 patients included at baseline.
Groups:
- Total: Total of all reporting groups
Arm/Group | SBRT for Benign Extradural Spine Tumors | SBRT for Vertebral/Paraspinal Metastases | Total
Number analyzed (Participants) | 3 | 35 | 38
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 2 | 20 | 22
  >=65 years | 1 | 15 | 16
Age, Continuous [Mean (Full Range); unit: years]
  Age Range | 64 [55 to 82] | 62 [34 to 90] | 62 [34 to 90]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 20 | 22
  Male | 1 | 15 | 16
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Race: Caucasion | 3 | 32 | 35
  Race: African American | 0 | 3 | 3
  Race: Other | 0 | 0 | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 3 | 35 | 38

OUTCOME MEASURES:

1. Primary Outcome: Initial Symptom Control
Description: Evaluation of pain relief per patient report
Time Frame: 6 weeks post-SBRT (or at first post-treatment follow-up)
Population: 2 enrolled pts were not treated. 35 pts completed 36 SBRT courses. 5 pts either died prior to any follow-up appointment or imaging (4 pts) or did not follow-up due to loss of insurance (1 pt). 3 pts with benign spine tumors and 28 pts with vertebral metastases who underwent a total of 32 courses of SBRT had follow-up data available for analysis.
Measure: Count of Participants; unit: Participants
Arm/Group | SBRT for Benign Extradural Spine Tumors | SBRT for Vertebral/Paraspinal Metastases
Number analyzed (Participants) | 3 | 28
Participants
  Number with Follow-up Data | 3 | 28
  Number with Initial Symptom Control | 3 | 27
  Number without Symptom Control | 0 | 1

2. Primary Outcome: Local Tumor Recurrence Rate
Description: Local recurrence is defined as tumor recurrence or progression within the planning target volume.
  Local control rate will be evaluated by imaging techniques and/or clinical symptoms (worsening or no improvement in pain or neurologic compromise). If follow-up imaging is available, a local recurrence will be defined as an increase of > 20% in tumor size.
Time Frame: (1) At 1 year post-SBRT, (2) At patient's last follow-up or time of death
Population: 35 pts completed 36 SBRT courses. All 3 benign tumor pts are still alive. 15 pts with metastatic disease died prior to first post-SBRT follow-up appointment or imaging (4 pts), did not follow-up due to loss of insurance (1 pt), or had initial follow-up but then died prior to 1 year from treatment completion (10 pts).
Measure: Count of Participants; unit: Participants
Arm/Group | SBRT for Benign Extradural Spine Tumors | SBRT for Vertebral/Paraspinal Metastases
Number analyzed (Participants) | 3 | 28
Participants
  Local Control at last Follow-up | 3 | 25
  No Response to Treatment | 0 | 1
  Local Recurrence after Initial Response | 0 | 2
  Number with at least 1 year Follow-up | 3 | 18
  Local Control at 1 year Follow-up | 3 | 17
  Local Recurrence within 1st year of Follow-up | 0 | 1

3. Secondary Outcome: Late Toxicity Rate
Description: Toxicity will be assessed using CTCAE grading criteria at specified timepoints.
Time Frame: at patient's last follow-up (at least 3 months from treatment) or time of death
Population: as for outcome 1
Measure: Number; unit: participants
Arm/Group | SBRT for Benign Extradural Spine Tumors | SBRT for Vertebral/Paraspinal Metastases
Number analyzed (Participants) | 3 | 28
participants | 0 | 0

ADVERSE EVENTS:
Time Frame: Patients were followed until time of death or until lost to follow-up.
Description: Serious adverse events are defined as events that result in either death, a life-threatening adverse event, inpatient hospitalization or prolongation of existing hospitalization, a persistent or significant incapacity or substantial disruption of the ability to conduct normal functions, or a congenital anomaly/birth defect. Events not meeting this definition are listed under Other Adverse Events (not serious). Only 28 of the patients within the metastases arm had follow-up data collected.
Arm/Group | SBRT for Benign Extradural Spine Tumors | SBRT for Vertebral/Paraspinal Metastases
All-Cause Mortality (participants affected / at risk) | 0/3 | 27/28
Serious Adverse Events (participants affected / at risk) | 0/3 | 1/28
Other Adverse Events (participants affected / at risk) | 1/3 | 7/28
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | SBRT for Benign Extradural Spine Tumors (N=3) | SBRT for Vertebral/Paraspinal Metastases (N=28)
Esophagitis (Gastrointestinal disorders) | 0 (0) | 1 (1) — Esophagitis requiring management with triple mix (Benadryl/Maalox/Lidocaine), oral steroids, Vicodin, and a soft diet, and resulted in < 10 pound weight loss.
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | SBRT for Benign Extradural Spine Tumors (N=3) | SBRT for Vertebral/Paraspinal Metastases (N=28)
Self limiting nausea (Gastrointestinal disorders) | 1 (1) | 3 (3)
desquamation (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) — skin redness and peeling
mild esophagitis (Gastrointestinal disorders) | 0 (0) | 2 (2) — esophagitis lasting less than 7 days, not interfering with eating, no or minimal intervention required
muscle pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) — temporary increased pain at treated site

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2013-02-04): https://cdn.clinicaltrials.gov/large-docs/07/NCT01347307/Prot_SAP_000.pdf